CLINICAL TRIAL: NCT05741190
Title: Correlation of Angle Kappa , Corneal High Order Aberrations and Total Eye Aberrations in Various Refractive Errors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mario Magdy Ezzat, Resident Doctor, Sohag University
Other Study IDs: Angle Kappa and aberrations
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-02

CONDITIONS: Aberration, Corneal Wavefront
MeSH Terms: conditions — Corneal Wavefront Aberration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- myope: Patients with myopia
  Interventions: Device: Pentacam Imaging
- Hypermetrope: Patients with hypermetropia
  Interventions: Device: Pentacam Imaging
- Astigmatic: Patients with Astigmatism
  Interventions: Device: Pentacam Imaging

INTERVENTIONS:
Device: Pentacam Imaging — Imaging of the corneal surface

SUMMARY:
Identification of the correlation between angle kappa , corneal high order aberrations and total eye aberrations in myopic hyperopic and astigmatic patients

DETAILED DESCRIPTION:
The patient will be thoroughly examined clinically on slit lamp detailed history will be obtained visual acuity will be measured and patient refraction will be taken then imaging on Sirius topographer will be used to obtain angle Kappa and high order aberrations of the cornea and I-design pentacam imaging will be used to get the total aberrations of the eye

ELIGIBILITY:
Inclusion Criteria:

1. Patients with errors of refraction above the age of 18
2. No history of trauma.
3. No other ocular disease .

Exclusion Criteria:

1. patient under age of 18
2. patients with systemic disease.
3. patient with corneal diseases
4. Patient who did any sort of occular surgery
5. patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with no ocular disease other than errors of refraction over 18 years old
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
correlation between angle Kappa and high order aberrations of the cornea and total aberrations of the eye in various refractive errors | baseline
  does the refraction affect the angle kappa or the corneal high order aberrations or the total aberrations of the eye

REFERENCES:
- [Background] Gharieb Ibrahim HM, Gharieb HM, Othman IS. Angle kappa Measurement and Its Correlation with Other Ocular Parameters in Normal Population by a New Imaging Modality. Optom Vis Sci. 2022 Jul 1;99(7):580-588. doi: 10.1097/OPX.0000000000001910. Epub 2022 Jun 3. PMID 35657347